CLINICAL TRIAL: NCT01592331
Title: A Single-Center, Randomized, Investigator/Subject-Blind, Single Dose, Placebo-Controlled, Parallel Group Study to Investigate the Pharmacodynamic and Pharmacokinetic Behavior of RO5508887 in Plasma and Cerebral Spinal Fluid Following Oral Administration in Healthy Volunteers
Brief Title: A Pharmacodynamic and Pharmacokinetic Study of RO5508887 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: WP27959
Record Dates: First submitted 2012-04-19; First posted 2012-05-07 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- RO5508887 (Experimental)
  Interventions: Drug: RO5508887

INTERVENTIONS:
Drug: Placebo — Single oral dose
  Arms: Placebo
Drug: RO5508887 — Single oral dose
  Arms: RO5508887

SUMMARY:
This randomized, double-blind, placebo-controlled, parallel group study will evaluate the pharmacodynamics and pharmacokinetics of RO5508887 in healthy volunteers.

Subjects will be randomized in cohorts to receive single oral doses of either RO5508887 or placebo. In-unit period is 6 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, 18 to 65 years of age, inclusive. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history and a complete physical examination
* Body mass index (BMI) 18 to 30 kg/m2 inclusive
* Must agree to use a barrier method of contraception during the treatment period and for at least 30 days after the last dose of study drug
* Donation of blood over 500 mL within 6 weeks before drug administration

Exclusion Criteria:

* Concomitant disease or condition or treatment that could interfere with the conduct of the study or would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
* Allergy to lidocaine
* Suspicion of regular consumption of drug of abuse
* Regular smoker (> 5 cigarettes, > 1 pipeful or > 1 cigar per day)
* Positive for hepatitis B, hepatitis C or HIV 1 or 2 infection
* Participation in an investigational drug or device study (last administration of study drug or installation of device) within 6 weeks before RO5508887 administration and within 5 mean half-lives of receiving previous investigational drug before RO5508887 administration. In addition, subject cannot participate unless completely recovered from previous invasive or study procedure
* Donation of blood over 500 mL within 6 weeks before drug administration

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Plasma levels of amyloid biomarkers | Pre-dose and up to fullow up, 8-12 days post dose
Cerebral spinal fluid levels of amyloid biomarkers | Pre-dose and up to 30 hours post-dose

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 6 months
Pharmacokinetics: Plasma and cerebral spinal fluid concentrations of RO5508887 (and metabolites) | Pre-dose and up to 72 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Glendale, California, United States